CLINICAL TRIAL: NCT02144493
Title: Case-control Study of Risk Factors for Recurrence of Primary Bile Duct Stones
Brief Title: Risk Factors for Recurrence of Primary Bile Duct Stones
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chuncheon Sacred Heart Hospital (Other)
Responsible Party: Principal Investigator, Jai Hoon Yoon, Professor Jai Hoon Yoon, Chuncheon Sacred Heart Hospital
Other Study IDs: YJH-1; ChuncheonSHH YJH-1 (Other: ChuncheonSHH)
Record Dates: First submitted 2014-05-12; First posted 2014-05-22 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Common Bile Duct Stones
Keywords: common bile duct stones; diverticulum
MeSH Terms: conditions — Diverticulum

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Patients with recurrent CBD stone
  Interventions: Other: The existence of periampullary diverticulum; Other: CBD angle
- Patients without recurrent CBD stone
  Interventions: Other: The existence of periampullary diverticulum; Other: CBD angle

INTERVENTIONS:
Other: The existence of periampullary diverticulum — Periampullary diverticulum has been postulated as risk factor of recurrent CBD stone.
Other: CBD angle — Narrow CBD angle has been postulated as risk factor for the development of recurrent CBD stone

SUMMARY:
Recurrent common bile duct stone is one of the risk factors of recurrent cholangitis. However, the exact pathophysiology or mechanism of recurrent cholangitis has not been established. Periampullary diverticulum and narrow angle of common bile duct have been postulated as risk factors of recurrent common bile duct stone. The aim of this study was to evaluate the association between periampullary dierticulum, angle of common bile duct and recurrent common bile duct stone.

DETAILED DESCRIPTION:
Recurrent common bile duct stone is one of the risk factors of recurrent cholangitis. However, the exact pathophysiology or mechanism of recurrent cholangitis has not been established. Periampullary diverticulum and narrow angle of common bile duct have been postulated as risk factors of recurrent common bile duct stone. The aim of this study was to evaluate the association between periampullary dierticulum, angle of common bile duct and recurrent common bile duct stone.

This study is patient-control setting study. Firstly, from July 2007 through February 2014, all the patients who were performed ERCP will be enrolled. The inclusion criteria is the patients with common bile duct stone. The exclusion criteria is patients with biliary stenosis, PSC, retained GB stone, or who were lost to follow-up. The main outcome is the association between periampullary diverticulum, common bile duct angle, and recurrent CBD stone. This will be evaluated by univariate and multivariate analyses.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were performed ERCP due to CBD stone or calculous cholangitis

Exclusion Criteria:

* Patients with biliary stricture, PSC, retained GB stone, or who were lost to follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed as CBD stone or calculous cholangitis will be enrolled. These patients will be divided by patienst with recurrent CBD stone (devlopment of CBD stone after 1 year from the first development of CBD stone) or not .
Sampling Method: Non-Probability Sample
Enrollment: 2 (Estimated)
Dates: Start 2014-05; Primary Completion 2014-12 (Estimated); Study Completion 2014-12 (Estimated)

PRIMARY OUTCOMES:
The association between existence of periampullary diverticulum and recurrent CBD stone | retrospective (up to 8 years)
  The association between existence of periampullary diverticulum and recurrent CBD stone will be assessed by univariate analysis.(unit of analysis: odds ratio, statistical method: Fisher's exact test)

SECONDARY OUTCOMES:
The association between common bile duct angle and existence of recurrent CBD stone | retrospective (up to 8 years)
  The association between common bile duct angle and recurrent CBD stone will be assessed by univariate analysis (unit of analysis: angle, statistical method: student's t test)

OTHER OUTCOMES:
The risk factors for the development of recurrent CBD stone | retrospective (up to 8 years)
  The risk factors for the development of recurrent CBD stone will be assessed by multivariate analysis, based on results of univariate analyses. (statistical method: logistic regression analysis)

CONTACTS AND LOCATIONS:
Overall Officials: Jai Hoon Yoon, M.D..Ph.D., Study Chair — Hallym University College of Medicine, Chuncheon Sacred Heart hospital
Locations (1):
- Chuncheon Sacred Heart Hospital, Chuncheon, Gangwon-do, South Korea

REFERENCES:
- [Background] Keizman D, Shalom MI, Konikoff FM. An angulated common bile duct predisposes to recurrent symptomatic bile duct stones after endoscopic stone extraction. Surg Endosc. 2006 Oct;20(10):1594-9. doi: 10.1007/s00464-005-0656-x. Epub 2006 Jul 20. PMID 16858527
- [Background] Katsinelos P, Chatzimavroudis G, Tziomalos K, Zavos C, Beltsis A, Lazaraki G, Terzoudis S, Kountouras J. Impact of periampullary diverticula on the outcome and fluoroscopy time in endoscopic retrograde cholangiopancreatography. Hepatobiliary Pancreat Dis Int. 2013 Aug;12(4):408-14. doi: 10.1016/s1499-3872(13)60063-6. PMID 23924499
- [Background] Panteris V, Vezakis A, Filippou G, Filippou D, Karamanolis D, Rizos S. Influence of juxtapapillary diverticula on the success or difficulty of cannulation and complication rate. Gastrointest Endosc. 2008 Nov;68(5):903-10. doi: 10.1016/j.gie.2008.03.1092. Epub 2008 Jul 16. PMID 18635174